CLINICAL TRIAL: NCT00578786
Title: A Long Term Study of Ambrisentan in Pulmonary Arterial Hypertension Subjects Having Completed AMB-320 (NCT00423748) or AMB-321 (NCT00423202)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMB-320/321-E; ARIES-E
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ambrisentan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ambrisentan (Experimental): 2.5, 5 or 10 mg ambrisentan
  Interventions: Drug: ambrisentan

INTERVENTIONS:
Drug: ambrisentan — 2.5, 5.0 or 10.0 mg ambrisentan po, qd, long-term
  Other Names: Letairis(TM)

SUMMARY:
AMB-320/321-E was designed to provide long-term, controlled monitoring of pulmonary arterial hypertension (PAH) patients treated with ambrisentan (AMB) in order to properly define the adverse event profile associated with this endothelin receptor antagonist (ERA), including the incidence and severity of elevated serum liver function tests (LFTs). In addition, this study continued the efficacy assessments of the previous studies, examined long-term AMB treatment success, and compared long-term survival of subjects treated with AMB to the NIH registry of patients with PAH.

DETAILED DESCRIPTION:
AMB-320 (ARIES-1; NCT00423748) and AMB-321 (ARIES-2; NCT00423202) were 12-week, Phase 3, randomized, double-blind, placebo-controlled, multicenter, efficacy studies of AMB in subjects with PAH. The objectives of these studies were to determine the effect of three doses of AMB (2.5, 5.0, and 10.0 mg) on exercise capacity, as well as several clinical measures of PAH. The current study (NCT00578786) was unblinded (by design) prior to completion. The ARIES studies were identical except for the dose groups assessed and the geographic locations where the studies were conducted. Both studies evaluated placebo and 5.0-mg AMB dose groups; however, AMB-320 (NCT00423748) also examined an AMB dose of 10.0 mg, while AMB-321 (NCT00423202) included an AMB dose of 2.5 mg. AMB-320/321-E was an optional study for subjects who had participated in AMB-320 (NCT00423748) or AMB-321 (NCT00423202) that allowed continued long-term treatment with AMB.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have completed Week 12 of AMB-320 (NCT00423748) or AMB-321 (NCT00423202) or must have received placebo during AMB-320 (NCT00423748) or AMB-321 (NCT00423202) and met two or more early escape criteria;
2. Subject must be competent to understand the information given in the Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approved informed consent form and must sign the form prior to the initiation of any study procedures.
3. Female subject of childbearing potential must agree to use two reliable methods of contraception until study completion and for at least four weeks following their final study visit. Reliable methods include: birth control pills/implants/injections, intrauterine devices (IUDs), spermicide, diaphragms, or condoms.

Exclusion Criteria:

* Subjects must have met the exclusion criteria of the AMB-320 (NCT00423748) and AMB-321 (NCT00423202)studies. In addition, a subject who meets any one of the following criteria is ineligible for participation in the study:

  1. Subject receiving bosentan, sildenafil, or iv inotropes at any time within four weeks prior to the AMB-320/321-E Screening/Randomization Visit;
  2. Subject receiving chronic prostanoid therapy (epoprostenol, treprostinil, iloprost, beraprost, or any other investigational prostacyclin derivative) within four weeks prior to the AMB-320/321-E Screening/RandomizationVisit;
  3. Female subject who is pregnant or breastfeeding;
  4. Subject with cardiovascular, liver, renal, hematologic, gastrointestinal, immunologic, endocrine, metabolic, or central nervous system disease that, in the opinion of the Investigator, may adversely affect the safety of the subject and/or efficacy of the study drug or severely limit the lifespan of the subject;
  5. Subject who has demonstrated noncompliance with previous medical regimens;
  6. Subject who has a recent history of abusing alcohol or illicit drugs;
  7. Subject who has participated in a clinical study involving another investigational drug or device at any time within four weeks prior to the AMB-320/321-E Screening/Randomization Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2004-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Dufton, PhD, Study Chair — Gilead Sciences
Locations (22):
- Argentina (11):
  - Sanatorio Otamendi, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Britanico-Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto del Corazon Denton A. Cooley, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - UAI Hosp. Universitario, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - HIGA Hospital Interzonal General de Agudos Oscar Allende, Mar del Plata, Buenos Aires
  - Clinica Independencia Munro, Munro, Buenos Aires
  - Instituto de Cardiologia J.F. Cabral, Corrientes, Corrientes Province
  - Sanatorio Allende, Córdoba, Córdoba Province
  - Hospital Italiano de Cordoba, Córdoba, Córdoba Province
  - Hospital Italiano de Rosario, Rosario, Sante Fe
  - Hospital Privado Centro Medico de Cordoba, Córdoba
- Brazil (6):
  - Hospital Universitario Clementino Fraga Filho, Ilha Do Fundao, Rio de Janeiro
  - Hospital Madre Teresa, Belo Horizonte
  - Hospital San Lucas de Pontificia Universidade Catolica, Porto Alegre
  - Complexo Hospitalar Sanata Casa de Porto Alegre, Porto Alegre
  - Universidade do Estado de Sao Paulo - UNIFESP, São Paulo
  - Hospital das Clinicas da FMUSP, São Paulo
- Chile (3):
  - Hospital San Juan de Dios, Santiago, Santiago de Chile
  - Hospital Clinico Universidad Catolica, Santiago, Santiago de Chile
  - Instituto Nacional del Torax, Santiago, Santiago de Chile
- Mexico (2):
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City, Mexico City
  - Unidad De Investigacion Clinica en Medicina, Monterrey, Nuevo Leon, Nuevo León

REFERENCES:
- [Derived] Oudiz RJ, Galie N, Olschewski H, Torres F, Frost A, Ghofrani HA, Badesch DB, McGoon MD, McLaughlin VV, Roecker EB, Harrison BC, Despain D, Dufton C, Rubin LJ; ARIES Study Group. Long-term ambrisentan therapy for the treatment of pulmonary arterial hypertension. J Am Coll Cardiol. 2009 Nov 17;54(21):1971-81. doi: 10.1016/j.jacc.2009.07.033. PMID 19909879

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants completing Week 12 of NCT00423748 or NCT00423202 could enroll in extension (E) study. Participants on placebo in parent study and d/c treatment due to >/=2 early escape criteria were eligible. Total randomized: 361 (completed/early escape in prior study), 19 (d/c prior study), and 3 (completed prior study, did not enroll in E study).
Pre-assignment Details: Participants on active treatment in NCT00423748 or NCT00423202 continued to receive their last assigned blinded ambrisentan (AMB) dose from the prior study. Those on placebo in NCT00423748 were randomized to receive either 5 or 10 mg of AMB in the extension study. Those on placebo in NCT00423202 were randomized to either 2.5 or 5 mg of AMB.
Groups:
- Ambrisentan 2.5 mg: Original randomized dose group in the prior study (NCT00423748 and NCT00423202) or in the current study (for subjects originally randomized to placebo in one of the prior studies). Analysis included those not enrolling in this study but received AMB in 1 of the 2 parent studies. It should be noted that by Year 3, almost half of those randomized to AMB 2.5 mg were titrated to 5 mg and 10 mg.
- Ambrisentan 5 mg: Original randomized dose group in the prior study (NCT00423748 and NCT00423202) or in the current study (for subjects originally randomized to placebo in one of the prior studies). Analysis included those not enrolling in this study but received AMB in 1 of the 2 parent studies. It should be noted that by Year 3, a third starting at 5 mg were titrated to 10 mg.
- Ambrisentan 10 mg: Original randomized dose group in the prior study (NCT00423748 and NCT00423202) or in the current study (for subjects originally randomized to placebo in one of the prior studies).
Period: Overall Study
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg
Started | 96 | 190 | 97
Completed | 57 | 124 | 67
Not Completed | 39 | 66 | 30
Not completed — Adverse Event | 27 | 37 | 17
Not completed — Lack of Efficacy | 2 | 5 | 2
Not completed — Early Escape from Prior Study | 2 | 1 | 2
Not completed — Withdrawal by Subject | 7 | 8 | 5
Not completed — Protocol Violation | 0 | 3 | 1
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Sponsor Decision | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 4 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Not Otherwise Specified | 0 | 4 | 1
Not completed — Qualified but Not Enrolled in Extension | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Total
Number analyzed (Participants) | 96 | 190 | 97 | 383
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline data values established at the screening/randomization visit of the 2 prior (parent) studies defined the baseline of this long-term analysis for subjects who first received 2.5, 5, or 10 mg ambrisentan in the prior studies. The Screening/Randomization Visit of the present extension study defined the baseline for subjects who received placebo in the 2 prior studies.
  years | 52.27 (14.968) | 51.46 (14.429) | 49.09 (16.572) | 51.06 (15.139)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 154 | 79 | 302
  Male | 27 | 36 | 18 | 81
Race/Ethnicity, Customized [Number; unit: participants] — Baseline data values established at the screening/randomization visit of the 2 prior (parent) studies defined the baseline of this long-term analysis for subjects who first received 2.5, 5, or 10 mg ambrisentan in the prior studies. The Screening/Randomization Visit of the present extension study defined the baseline for subjects who received placebo in the 2 prior studies.
  participants
    Caucasian | 81 | 148 | 65 | 294
    Black | 0 | 5 | 6 | 11
    Asian | 1 | 6 | 2 | 9
    Hispanic | 14 | 29 | 22 | 65
    Other | 0 | 2 | 2 | 4
Pulmonary Arterial Hypertension Stratification [Number; unit: participants] — Participants were classified as diagnosed with idiopathic pulmonary arterial hypertension (IPAH) or non-idiopathic PAH (non-IPAH). Baseline data values established at the screening/randomization visit of the 2 prior (parent) studies defined the baseline of this long-term analysis for subjects who first received 2.5, 5, or 10 mg ambrisentan in the prior studies. The Screening/Randomization Visit of the present extension study defined the baseline for subjects who received placebo in the 2 prior studies.
  participants
    Idiopathic PAH (IPAH) | 63 | 119 | 59 | 241
    Non-IPAH | 33 | 71 | 38 | 142
6-Minute Walk Distance (6MWD) [Mean (Standard Deviation); unit: meters] — A measure of the distance participants could walk in 6 minutes. Baseline data values established at the screening/randomization visit of the 2 prior (parent) studies defined the baseline of this long-term analysis for subjects who first received 2.5, 5, or 10 mg ambrisentan in the prior studies. The Screening/Randomization Visit of the present extension study defined the baseline for subjects who received placebo in the 2 prior studies.
  meters | 350.3 (86.640) | 347.7 (87.333) | 342.3 (80.840) | 347.0 (85.389)
World Heath Organization (WHO) Class [Number; unit: participants] — WHO Classes: I) pulmonary hypertension (PH); ordinary physical activity not limited or causes increased dyspnea, fatigue, chest pain, or presyncope. II) PH; ordinary physical activity mildly limits/causes increased dyspnea, fatigue, chest pain, or presyncope; comfortable at rest. III) PH; physical activity markedly limited and less than ordinary physical activity causes increased dyspnea, fatigue, chest pain, or presyncope; comfortable at rest. IV) PH; physical activity causes symptoms; signs of right heart failure; dyspnea/fatigue possible at rest. Baseline defined as previously described.
  participants
    WHO Class I | 1 | 7 | 4 | 12
    WHO Class II | 51 | 77 | 35 | 163
    WHO Class III | 39 | 91 | 48 | 178
    WHO Class IV | 5 | 15 | 10 | 30
Borg Dyspnea Index (BDI) [Mean (Standard Deviation); unit: units on a scale] — Borg Dyspnea Index is a measure of perceived shortness of breath: 0 units on a scale (none) to 10 units on a scale (maximum breathlessness). Baseline data values established at the screening/randomization visit of the 2 prior (parent) studies defined the baseline of this long-term analysis for subjects who first received 2.5, 5, or 10 mg ambrisentan in the prior studies. The Screening/Randomization Visit of the present extension study defined the baseline for subjects who received placebo in the 2 prior studies.
  units on a scale | 4.14 (2.684) | 3.80 (2.332) | 3.78 (2.133) | 3.88 (2.377)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Adult body mass index (BMI) is calculated by dividing weight in kg by height in meters squared.BMI below 18.5 = underweight; BMI 18.5 to 24.9 = normal; BMI 25.0 to 29.9 = overweight; BMI 30.0 and above = obese. Note that 1 subject was not included in the denominator for the Ambrisentan 5 mg group (N=189) and the combined group (N=382). Baseline was defined as previously described.
  kg/m^2 | 26.68 (5.038) | 26.86 (5.632) | 28.26 (7.212) | 27.17 (5.958)

OUTCOME MEASURES:

1. Secondary Outcome: Baseline Exercise Capacity as Measured by the 6-Minute Walk Distance Test
Description: The 6-minute walk distance (6MWD) test was conducted according to the American Thoracic Society guidelines (ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med 2002; 166(1):111-117.).
Time Frame: Baseline
Population: All assessments of efficacy were performed using the randomized analysis set; subjects were allotted to an individual dose group based upon their randomized treatment assignment in the 2 prior studies (NCT00423748 or NCT00423202) or in the extension study. The LOCF method of imputation was used; only postbaseline observations were carried forward.
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- Ambrisentan 2.5 mg; Ambrisentan 5 mg; Ambrisentan 10 mg: Participants were classified based on their randomized dose of AMB in the 2 prior studies (NCT00423748 or NCT00423202) or in the current extension study. Study drug was taken once daily.
- Combined Ambrisentan Group: All dose groups combined.
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Combined Ambrisentan Group
Number analyzed (Participants) | 96 | 190 | 97 | 383
Meters | 350.3 (86.64) | 347.7 (87.33) | 342.3 (80.84) | 347.0 (85.39)

2. Primary Outcome: Frequently Reported (15% or More Overall) Adverse Events by Severity
Description: The primary endpoint of this study is the incidence and severity of adverse events associated with long-term exposure to AMB in participants with PAH. The most frequently occurring adverse events (occurring in 15% or more of the participants in the combined group) are presented, by severity, that began after entering this extension study. Adverse events that were serious are included. Adverse events are coded according to the Medical Dictionary for Regulatory Activities (MedDRA) Version 6.1 and are presented by MedDRA preferred term. Severity was graded as follows: mild (AE did not interfere with routine activities; subject may have experienced slight discomfort), moderate (AE interfered with routine activities; subject may have experienced significant discomfort), and severe (AE made it impossible to perform routine activities; subject may have experienced intolerable discomfort or pain).
Time Frame: Baseline to Week 295
Population: Safety Analysis Set: Includes all participants who received at least 1 dose of AMB in one of the 2 prior studies (NCT00423748 or NCT00423202) or in the current extension study. Treatment group assignments for the safety analysis set were based upon the highest dose of AMB received at any time during the parent or extension studies.
Measure: Number; unit: participants
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg
Number analyzed (Participants) | 43 | 146 | 194
participants
  Headache - Mild | 1 | 20 | 36
  Headache - Moderate | 0 | 14 | 17
  Headache - Severe | 0 | 0 | 8
  Pulmonary hypertension (worsening) - Mild | 2 | 2 | 7
  Pulmonary hypertension (worsening) - Moderate | 4 | 10 | 29
  Pulmonary hypertension (worsening) - Severe | 6 | 6 | 19
  Right ventricular failure - Mild | 0 | 2 | 6
  Right ventricular failure - Moderate | 2 | 7 | 14
  Right ventricular failure - Severe | 5 | 12 | 26
  Cough - Mild | 1 | 23 | 24
  Cough - Moderate | 1 | 2 | 22
  Cough - Severe | 0 | 1 | 0
  Upper respiratory tract infection - Mild | 3 | 13 | 23
  Upper respiratory tract infection - Moderate | 2 | 4 | 26
  Upper respiratory tract infection - Severe | 0 | 0 | 1
  Dizziness - Mild | 1 | 8 | 31
  Dizziness - Moderate | 2 | 7 | 14
  Dizziness - Severe | 0 | 0 | 3
  Dyspnoea exacerbated - Mild | 1 | 4 | 8
  Dyspnoea exacerbated - Moderate | 3 | 14 | 22
  Dyspnoea exacerbated - Severe | 1 | 2 | 7
  Arthralgia - Mild | 1 | 5 | 19
  Arthralgia - Moderate | 3 | 11 | 18
  Arthralgia - Severe | 1 | 2 | 1
  Diarrhoea - Mild | 2 | 12 | 17
  Diarrhoea - Moderate | 1 | 10 | 15
  Diarrhoea - Severe | 0 | 2 | 1
  Nasopharyngitis - Mild | 1 | 14 | 19
  Nasopharyngitis - Moderate | 1 | 8 | 15
  Nasopharyngitis - Severe | 0 | 0 | 0
  Oedema peripheral - Mild | 6 | 31 | 48
  Oedema peripheral - Moderate | 6 | 19 | 50
  Oedema peripheral - Severe | 1 | 3 | 4

3. Secondary Outcome: Change From Baseline to Week 24 in Exercise Capacity as Measured by the 6-Minute Walk Distance Test
Description: The 6-minute walk distance (6MWD) test was conducted according to the American Thoracic Society guidelines (ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med 2002; 166(1):111-117.). Missing values were imputed using LOCF method based on post-baseline observations. Baseline (BL) values from the screening/randomization visit of the 2 prior studies defined the BL of this long-term analysis for those receiving ambrisentan in the prior studies. The Screening/Randomization Visit of the present study was the BL for subjects receiving placebo in the prior studies.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- Ambrisentan 2.5 mg; Ambrisentan 5 mg; Ambrisentan 10 mg: Participants were classified based on their randomized dose of ambrisentan in the 2 prior studies (NCT00423748 or NCT00423202) or in the current extension study. Study drug was taken once daily.
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Combined Ambrisentan Group
Number analyzed (Participants) | 93 | 186 | 96 | 375
Meters | 38.0 (74.28) | 32.5 (78.55) | 40.9 (72.85) | 36.0 (75.97)
Statistical Analysis 1: Comparison: Ambrisentan 2.5 mg; Test type: Superiority or Other; Mean Difference (Net) = 38.0, 95% CI 2-sided [22.7 to 53.3], Standard Deviation 74.28 — Applies to Ambrisentan 2.5 mg group only. Missing values were imputed using last-observation-carried forward method (LOCF) based on post-baseline observations
Statistical Analysis 2: Comparison: Ambrisentan 5 mg; Test type: Superiority or Other; Mean Difference (Net) = 32.5, 95% CI 2-sided [21.1 to 43.8], Standard Deviation 78.55 — Applies to Ambrisentan 5 mg group only. Missing values were imputed using last-observation-carried forward method (LOCF) based on post-baseline observations
Statistical Analysis 3: Comparison: Ambrisentan 10 mg; Test type: Superiority or Other; Mean Difference (Net) = 40.9, 95% CI 2-sided [26.1 to 55.7], Standard Deviation 72.85 — Applies to Ambrisentan 10 mg group only. LOCF method of imputation. Missing values were imputed using last-observation-carried forward method (LOCF) based on post-baseline observations
Statistical Analysis 4: Comparison: Combined Ambrisentan Group; Test type: Superiority or Other; Mean Difference (Net) = 36.0, 95% CI 2-sided [28.3 to 43.7], Standard Deviation 75.97 — Applies to Ambrisentan combined group only. LOCF method of imputation

4. Secondary Outcome: Change From Baseline to Week 48 (Year 1) in Exercise Capacity as Measured by the 6-Minute Walk Distance Test
Description: The 6-minute walk distance (6MWD) test was conducted according to the American Thoracic Society guidelines (ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med 2002; 166(1):111-117.). The last-observation-carried-forward (LOCF) imputation method was used. Baseline (BL) values from the screening/randomization visit of the 2 prior studies defined the BL of this long-term analysis for those receiving AMB in the prior studies. The Screening/Randomization Visit of the present study was the BL for subjects receiving placebo in the prior studies.
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- Ambrisentan Combined Group: All dose groups combined.
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Ambrisentan Combined Group
Number analyzed (Participants) | 93 | 186 | 96 | 375
Meters | 24.9 (96.14) | 27.9 (94.50) | 37.2 (72.97) | 29.5 (89.81)
Statistical Analysis 1: Comparison: Ambrisentan 2.5 mg; Test type: Superiority or Other; Mean Difference (Net) = 24.9, 95% CI 2-sided [5.1 to 44.7], Standard Deviation 96.14 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Ambrisentan 5 mg; Test type: Superiority or Other; Mean Difference (Net) = 27.9, 95% CI 2-sided [14.2 to 41.6], Standard Deviation 94.50 — Applies to Ambrisentan 5.0 mg group only. Missing values were imputed using last-observation-carried forward method (LOCF) based on post-baseline observations
Statistical Analysis 3: Comparison: Ambrisentan 10 mg; Test type: Superiority or Other; Mean Difference (Net) = 37.2, 95% CI 2-sided [22.4 to 52.0], Standard Deviation 72.97 — Applies to Ambrisentan 10 mg group only. Missing values were imputed using last-observation-carried forward method (LOCF) based on post-baseline observations
Statistical Analysis 4: Comparison: Ambrisentan Combined Group; Test type: Superiority or Other; Median Difference (Net) = 29.5, 95% CI 2-sided [20.4 to 38.7], Standard Deviation 89.81 — Applies to Ambrisentan combined group only. LOCF method of imputation

5. Secondary Outcome: Change From Baseline to Year 2 in Exercise Capacity as Measured by the 6-Minute Walk Distance Test
Description: as for outcome 4
Time Frame: Baseline to Year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Combined Ambrisentan Group
Number analyzed (Participants) | 93 | 186 | 96 | 375
Meters | 6.7 (97.48) | 23.2 (100.69) | 28.0 (84.38) | 20.3 (96.05)
Statistical Analysis 1: Comparison: Ambrisentan 2.5 mg; Test type: Superiority or Other; Mean Difference (Net) = 6.7, 95% CI 2-sided [-13.4 to 26.8], Standard Deviation 97.48 — Applies to Ambrisentan 2.5 mg group only. LOCF method of imputation
Statistical Analysis 2: Comparison: Ambrisentan 5 mg; Test type: Superiority or Other; Mean Difference (Net) = 23.2, 95% CI 2-sided [8.7 to 37.8], Standard Deviation 100.69 — Applies to Ambrisentan 5 mg group only. LOCF method of imputation
Statistical Analysis 3: Comparison: Ambrisentan 10 mg; Test type: Superiority or Other; Mean Difference (Net) = 28.0, 95% CI 2-sided [10.9 to 45.1], Standard Deviation 84.38 — Applies to Ambrisentan 10 mg group only. LOCF method of imputation
Statistical Analysis 4: Comparison: Combined Ambrisentan Group; Test type: Superiority or Other; Median Difference (Net) = 20.3, 95% CI 2-sided [10.6 to 30.1], Standard Deviation 96.05 — Applies to Ambrisentan combined group only. Missing values were imputed using last-observation-carried forward method (LOCF) based on post-baseline observations

6. Secondary Outcome: Change From Baseline to Year 3 in Exercise Capacity as Measured by the 6-Minute Walk Distance Test
Description: Thoracic Society guidelines (ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med 2002; 166(1):111-117.). The last-observation-carried-forward (LOCF) imputation method was used. Baseline (BL) values from the screening/randomization visit of the 2 prior studies defined the BL of this long-term analysis for those receiving AMB in the prior studies. The Screening/Randomization Visit of the present study was the BL for subjects receiving placebo in the prior studies.
Time Frame: Baseline to Year 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Combined Ambrisentan Group
Number analyzed (Participants) | 93 | 186 | 96 | 375
Meters | 0.7 (95.21) | 18.8 (101.22) | 27.8 (87.07) | 16.6 (96.54)
Statistical Analysis 1: Comparison: Ambrisentan 2.5 mg; Test type: Superiority or Other; Mean Difference (Net) = 0.7, 95% CI 2-sided [-18.9 to 20.3], Standard Deviation 95.21 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Ambrisentan 5 mg; Test type: Superiority or Other; Mean Difference (Net) = 18.8, 95% CI 2-sided [4.2 to 33.5], Standard Deviation 101.22 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Ambrisentan 10 mg; Test type: Superiority or Other; Mean Difference (Net) = 27.8, 95% CI 2-sided [10.1 to 45.4], Standard Deviation 87.07 — [estimate comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Combined Ambrisentan Group; Test type: Superiority or Other; Mean Difference (Net) = 16.6, 95% CI 2-sided [6.8 to 26.4], Standard Deviation 96.54 — [estimate comment as in outcome 5, analysis 4]

7. Secondary Outcome: Baseline Borg Dyspnea Index
Description: Borg Dyspnea Index is a measure of perceived shortness of breath: 0 units on a scale (none) to 10 units on a scale (maximum breathlessness).
Time Frame: Baseline
Population: All assessments of efficacy were performed using the randomized analysis set, such that subjects were allotted to an individual dose group based upon their randomized treatment assignment in the 2 prior studies (NCT00423748 or NCT00423202) or in the current extension study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Combined Ambrisentan Group
Number analyzed (Participants) | 96 | 189 | 97 | 382
units on a scale | 4.14 (2.684) | 3.80 (2.332) | 3.78 (2.133) | 3.88 (2.377)

8. Secondary Outcome: Change From Baseline to Year 1 in Borg Dyspnea Index
Description: Borg Dyspnea Index is a measure of perceived shortness of breath: 0 units on a scale (none) to 10 units on a scale (maximum breathlessness). Baseline (BL) values from the screening/randomization visit of the 2 prior studies defined the BL of this long-term analysis for those receiving ambrisentan in the prior studies. The Screening/Randomization Visit of the present study was the BL for subjects receiving placebo in the prior studies.
Time Frame: Baseline to Year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Combined Ambrisentan Group
Number analyzed (Participants) | 93 | 185 | 96 | 374
units on a scale | -0.08 (2.254) | -0.59 (2.450) | -0.51 (2.400) | -0.44 (2.393)
Statistical Analysis 1: Comparison: Ambrisentan 2.5 mg; Test type: Superiority or Other; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.55 to 0.38], Standard Deviation 2.254 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Ambrisentan 5 mg; Test type: Superiority or Other; Mean Difference (Net) = -0.59, 95% CI 2-sided [-0.94 to -0.23], Standard Deviation 2.450 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Ambrisentan 10 mg; Test type: Superiority or Other; Mean Difference (Net) = -0.51, 95% CI 2-sided [-1.00 to -0.03], Standard Deviation 2.400 — [estimate comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Combined Ambrisentan Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.69 to -0.20], Standard Deviation 2.393 — [estimate comment as in outcome 5, analysis 4]

9. Secondary Outcome: Change From Baseline to Year 2 in Borg Dyspnea Index
Description: Borg Dyspnea Index is a measure of perceived shortness of breath: 0 units on a scale (none) to 10 units on a scale (maximum breathlessness). Baseline (BL) values from the screening/randomization visit of the 2 prior studies defined the BL of this long-term analysis for those receiving AMB in the prior studies. The Screening/Randomization Visit of the present study was the BL for subjects receiving placebo in the prior studies.
Time Frame: Baseline to Year 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Combined Ambrisentan Group
Number analyzed (Participants) | 93 | 185 | 96 | 374
units on a scale | 0.23 (2.603) | -0.33 (2.477) | -0.65 (2.305) | -0.27 (2.480)
Statistical Analysis 1: Comparison: Ambrisentan 2.5 mg; Test type: Superiority or Other; Mean Difference (Net) = 0.23, 95% CI 2-sided [-0.31 to 0.76], Standard Deviation 2.603 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Ambrisentan 5 mg; Test type: Superiority or Other; Mean Difference (Net) = -0.33, 95% CI 2-sided [-0.68 to 0.03], Standard Deviation 2.477 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Ambrisentan 10 mg; Test type: Superiority or Other; Mean Difference (Net) = -0.65, 95% CI 2-sided [-1.12 to -0.18], Standard Deviation 2.305 — [estimate comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Combined Ambrisentan Group; Test type: Superiority or Other; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.52 to -0.02], Standard Deviation 2.480 — [estimate comment as in outcome 5, analysis 4]

10. Secondary Outcome: Change From Baseline to Year 3 in Borg Dyspnea Index
Description: as for outcome 9
Time Frame: Baseline to Year 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Combined Ambrisentan Group
Number analyzed (Participants) | 93 | 185 | 96 | 374
units on a scale | 0.20 (2.593) | -0.14 (2.514) | -0.48 (2.215) | -0.14 (2.467)
Statistical Analysis 1: Comparison: Ambrisentan 2.5 mg; Test type: Superiority or Other; Mean Difference (Net) = 0.20, 95% CI 2-sided [-0.33 to 0.74], Standard Deviation 2.593 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Ambrisentan 5 mg; Test type: Superiority or Other; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.51 to 0.22], Standard Deviation 2.514 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Ambrisentan 10 mg; Test type: Superiority or Other; Mean Difference (Net) = -0.48, 95% CI 2-sided [-0.93 to -0.03], Standard Deviation 2.215 — [estimate comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Combined Ambrisentan Group; Test type: Superiority or Other; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.39 to 0.11], Standard Deviation 2.467 — [estimate comment as in outcome 5, analysis 4]

11. Secondary Outcome: Baseline World Health Organization (WHO) Functional Class
Description: WHO Classes: I) pulmonary hypertension (PH); ordinary physical activity not limited or causes increased dyspnea, fatigue, chest pain, or presyncope. II) PH; ordinary physical activity mildly limited and causes increased dyspnea, fatigue, chest pain, or presyncope; comfortable at rest. III) PH; physical activity markedly limited and less than ordinary physical activity causes increased dyspnea, fatigue, chest pain, or presyncope; comfortable at rest. IV) PH; physical activity causes symptoms; signs of right heart failure; dyspnea/fatigue possible at rest.
Time Frame: Baseline
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Ambrisentan Combined Group
Number analyzed (Participants) | 96 | 190 | 97 | 383
participants
  WHO Functional Class I | 1 | 7 | 4 | 12
  WHO Functional Class II | 51 | 77 | 35 | 163
  WHO Functional Class III | 39 | 91 | 48 | 178
  WHO Functional Class IV | 5 | 15 | 10 | 30

12. Secondary Outcome: Change From Baseline to Year 1 in World Health Organization (WHO) Functional Class
Description: as for outcome 11
Time Frame: Baseline to Year 1
Population: All assessments of efficacy were performed using the randomized analysis set; subjects were allotted to an individual dose group based upon their randomized treatment assignment in the 2 prior studies (NCT00423748 or NCT00423202) or in extension study. Missing values imputed using LOCF based on post-baseline observations.
Measure: Number; unit: participants
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Ambrisentan Combined Group
Number analyzed (Participants) | 96 | 190 | 97 | 383
participants
  Improved | 16 | 56 | 36 | 108
  No Change | 68 | 122 | 46 | 236
  Deteriorated | 10 | 9 | 14 | 33
  Missing | 2 | 3 | 1 | 6

13. Secondary Outcome: Change From Baseline to Year 2 in World Health Organization (WHO) Functional Class
Description: as for outcome 11
Time Frame: Baseline to Year 2
Population: All assessments of efficacy were performed using the randomized analysis set; subjects were allotted to an individual dose group based upon their randomized treatment assignment in the 2 prior studies (NCT00423748 or NCT00423202) or in extension study. Missing values were imputed using LOCF based on post-baseline observations.
Measure: Number; unit: participants
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Combined Ambrisentan Group
Number analyzed (Participants) | 96 | 190 | 97 | 383
participants
  Improved | 16 | 58 | 39 | 113
  No Change | 58 | 109 | 43 | 210
  Deteriorated | 20 | 20 | 14 | 54
  Missing | 2 | 3 | 1 | 6

14. Secondary Outcome: Change From Baseline to Year 3 in World Health Organization (WHO) Functional Class
Description: as for outcome 11
Time Frame: Baseline to Year 3
Population: All assessments of efficacy were performed using the randomized analysis set; subjects were allotted to an individual dose group based upon their randomized treatment assignment in the 2 prior studies (NCT00423748 or NCT00423202) or in the extension study. Missing values were imputed using LOCF based on post-baseline observations.
Measure: Number; unit: participants
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Combined Ambrisentan Group
Number analyzed (Participants) | 96 | 190 | 97 | 383
participants
  Improved | 17 | 61 | 32 | 110
  No Change | 57 | 109 | 49 | 215
  Deteriorated | 20 | 17 | 15 | 52
  Missing | 2 | 3 | 1 | 6

15. Secondary Outcome: Baseline SF-36 Health Survey Scales for the Combined Ambrisentan Group
Description: The 8 scales of the SF-36 Health Survey measured included physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health, and the summary measures included physical health and mental health. Scores for each scale are transformed and the transformed scores range from 0 (worst health) to 100 (best health). The scores are then standardized with the 1998 General United States (US) population mean and standard deviation (SD). Finally, the scores are transformed to the norm-based scoring with a mean of 50 and SD of 10.
Time Frame: Baseline
Population: All participants were combined into one group for this analysis (all doses) and an observed-case approach was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Ambrisentan Group
Number analyzed (Participants) | 355
units on a scale
  Physical Functioning | 30.0 (9.02)
  Role Physical | 35.2 (10.21)
  Bodily Pain | 46.3 (11.93)
  General Health | 36.0 (8.65)
  Vitality | 42.1 (10.23)
  Social Functioning | 39.6 (11.8)
  Role Emotional | 39.2 (13.47)
  Mental Health | 43.3 (12.12)
  Physical Component Summary | 35.1 (8.52)
  Mental Component Summary | 44.5 (11.98)

16. Secondary Outcome: Change From Baseline to Week 12 in SF-36 Health Survey Scales for the Combined Ambrisentan Group
Description: The 8 scales of the SF-36 Health Survey measured included physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health, and the summary measures included physical health and mental health. Scores for each scale are transformed and the transformed scores range from 0 (worst health) to 100 (best health). The scores are then standardized with the 1998 General US population mean and SD. Finally, the scores are transformed to the norm-based scoring with a mean of 50 and SD of 10.
Time Frame: Baseline to Week 12
Population: All participants were combined into one group for this analysis (all doses) and an observed-case approach was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Ambrisentan Group
Number analyzed (Participants) | 303
units on a scale
  Physical Functioning (n=299) | 3.9 (7.40)
  Role Physical (n=298) | 5.6 (10.81)
  Bodily Pain (n=303) | 1.8 (11.27)
  General Health (n=297) | 3.1 (7.85)
  Vitality (n=301) | 4.6 (9.12)
  Social Functioning (n=303) | 3.9 (10.63)
  Role Emotional (n=286) | 3.9 (14.69)
  Mental Health (n=301) | 3.2 (9.72)
  Physical Component Summary (n=276) | 3.8 (7.59)
  Mental Component Summary (n=276) | 3.4 (10.77)

17. Secondary Outcome: Change From Baseline to Week 24 in SF-36 Health Survey Scales for the Combined Ambrisentan Group
Description: as for outcome 16
Time Frame: Baseline to Week 24
Population: All participants were combined into one group for this analysis (all doses) and an observed-case approach was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Combined Ambrisentan Group: (All Doses)
Arm/Group | Combined Ambrisentan Group
Number analyzed (Participants) | 230
units on a scale
  Physical Functioning (n=226) | 4.7 (8.75)
  Role Physical (n=227) | 5.7 (13.37)
  Bodily Pain (n=230) | 1.0 (13.28)
  General Health (n=223) | 3.2 (8.11)
  Vitality (n=227) | 4.5 (9.55)
  Social Functioning (n=230) | 3.5 (11.50)
  Role Emotional (n=220) | 4.3 (14.45)
  Mental Health (n=227) | 2.6 (10.57)
  Physical Component Summary (n=212) | 3.8 (9.06)
  Mental Component Summary (n=212) | 3.2 (11.06)

18. Secondary Outcome: Change From Baseline to Week 36 in SF-36 Health Survey Scales for the Combined Ambrisentan Group
Description: as for outcome 16
Time Frame: Baseline to Week 36
Population: All participants were combined into one group for this analysis (all doses) and an observed-case approach was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Ambrisentan Group
Number analyzed (Participants) | 186
units on a scale
  Physical Functioning (n=183) | 4.9 (8.27)
  Role Physical (n=181) | 4.5 (12.34)
  Bodily Pain (n=186) | 1.9 (13.16)
  General Health (n=181) | 4.5 (12.34)
  Vitality (n=185) | 4.6 (9.16)
  Social Functioning (n=186) | 3.7 (12.26)
  Role Emotional (n=178) | 3.6 (15.17)
  Mental Health (n=185) | 2.9 (11.00)
  Physical Component Summary (n=169) | 3.9 (8.79)
  Mental Component Summary (n=169) | 2.9 (11.34)

19. Secondary Outcome: Percentage of Participants With No Clinical Worsening of PAH
Description: Clinical worsening of PAH was defined as the time from randomization to ambrisentan therapy to the first occurrence of death, lung transplantation, hospitalization for PAH, atrial septostomy, addition of approved prostanoid therapy, study withdrawal due to the addition of other clinically approved PAH therapeutics, or study withdrawal due to 2 or more early escape criteria (for subjects randomized to AMB in NCT00423748 or NCT00423202). Results are presented as the Kaplan-Meier estimate (% probability) of not having clinical worsening after a given time.
Time Frame: Baseline to Year 3
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percent probability (KM estimate)
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Ambrisentan Combined Group
Number analyzed (Participants) | 96 | 190 | 97 | 383
percent probability (KM estimate)
  No clinical worsening after 1 year of treatment | 80.4 (4.2) [70.7 to 87.2] | 83.9 (2.7) [77.7 to 88.5] | 82.8 (3.9) [73.5 to 89.1] | 82.7 (2.0) [78.4 to 86.2]
  No clinical worsening after 2 years of treatment | 67.8 (4.9) [57.0 to 76.4] | 72.4 (3.4) [65.1 to 78.5] | 72.2 (4.8) [61.7 to 80.3] | 71.1 (2.4) [66.1 to 75.6]
  No clinical worsening after 3 years of treatment | 60.7 (5.2) [49.7 to 70.0] | 67.4 (3.7) [59.7 to 74.0] | 59.9 (5.6) [48.0 to 69.9] | 63.8 (2.7) [58.4 to 68.8]

20. Secondary Outcome: Percentage of Participants With Failure-Free Treatment Status
Description: Treatment failure was defined as the time from randomization to ambrisentan therapy to the first occurrence of death, lung transplantation, addition of approved prostanoid therapy, study withdrawal due to the addition of other clinically approved PAH therapeutics, or study withdrawal due to 2 or more early escape criteria (for subjects randomized to ambrisentan in NCT00423748 or NCT00423202). Results are presented as the Kaplan-Meier estimate (% probability) of not having treatment failure after a given time.
Time Frame: Baseline to Year 4
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percent probability (KM estimate)
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Ambrisentan Combined Group
Number analyzed (Participants) | 96 | 190 | 97 | 383
percent probability (KM estimate)
  No treatment failure after 1 year of treatment | 86.8 (3.6) [77.9 to 92.3] | 89.0 (2.4) [83.3 to 92.9] | 90.1 (3.1) [81.8 to 94.7] | 88.7 (1.7) [85.0 to 91.6]
  No treatment failure after 2 years of treatment | 77.6 (4.4) [67.4 to 84.9] | 79.8 (3.1) [72.8 to 85.1] | 81.4 (4.2) [71.4 to 88.2] | 79.6 (2.2) [75.0 to 83.5]
  No treatment failure after 3 years of treatment | 69.1 (5.0) [58.3 to 77.7] | 73.8 (3.5) [66.2 to 80.0] | 67.9 (5.7) [55.5 to 77.6] | 71.3 (2.6) [65.9 to 76.0]
  No treatment failure after 4 years of treatment | 60.8 (5.4) [49.4 to 70.5] | 69.0 (4.0) [60.3 to 76.2] | 63.2 (6.2) [49.9 to 73.9] | 66.4 (2.8) [59.0 to 70.4]

21. Secondary Outcome: Long-term Survival
Description: Long-term survival was defined as the time from initiation of active treatment to death. Results are presented as the Kaplan-Meier estimate (% probability) of survival after a given time.
Time Frame: Baseline to Year 4
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percent probability (KM estimate)
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg | Ambrisentan Combined Group
Number analyzed (Participants) | 96 | 190 | 97 | 383
percent probability (KM estimate)
  Survival after 1 year of treatment | 96.8 (1.8) [90.4 to 99.0] | 93.1 (1.9) [88.1 to 96.0] | 94.5 (2.4) [87.2 to 97.7] | 94.4 (1.2) [91.4 to 96.3]
  Survival after 2 years of treatment | 84.7 (3.9) [75.1 to 90.8] | 87.3 (2.6) [81.2 to 91.6] | 90.7 (3.1) [82.3 to 95.3] | 87.5 (1.8) [83.5 to 90.6]
  Survival after 3 years of treatment | 78.4 (4.5) [67.9 to 85.8] | 84.2 (2.9) [77.4 to 89.1] | 82.7 (4.5) [71.7 to 89.7] | 82.2 (2.2) [77.5 to 86.1]
  Survival After 4 Years of Treatment | 71.1 (5.2) [59.6 to 79.9] | 78.1 (3.8) [69.5 to 84.6] | 82.7 (4.5) [71.7 to 89.7] | 76.5 (2.7) [70.7 to 81.3]

22. Primary Outcome: Serum Aminotransferases Relative to the Upper Limit of the Normal Range (ULN)
Description: The number of participants with serum alanine aminotransferase (ALT) and serum aspartate aminotransferase (AST) falling into the following categories: >3.0 and </= 5.0 x ULN, >5.0 and </= 8.0 x ULN, and >8.0 x ULN. Includes the highest value per participant across all visits as well as values from early termination visits.
Time Frame: Baseline to Week 295
Population: Safety Analysis Set: Includes all participants who received at least 1 blinded dose of AMB in one of the 2 prior studies (NCT00423748 or NCT00423202) or in the current extension study.
Measure: Number; unit: participants
Groups:
- Ambrisentan 2.5 mg; Ambrisentan 5 mg; Ambrisentan 10 mg: Participants were classified based on the highest dose of AMB received at any time during the 2 prior studies (NCT00423748 or NCT00423202) or in the current extension study. Study drug was taken once daily.
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg
Number analyzed (Participants) | 43 | 155 | 205
participants
  ALT >3.0 and </=5.0 x ULN | 0 | 2 | 4
  ALT >5.0 and </= 8.0 x ULN | 0 | 1 | 0
  ALT >8.0 x ULN | 0 | 3 | 5
  Total ALT results >3.0 x ULN | 0 | 0 | 1
  AST >3.0 and </=5.0 x ULN | 1 | 3 | 7
  AST >5.0 and </= 8.0 x ULN | 0 | 1 | 0
  AST >8.0 x ULN | 0 | 0 | 1
  Total AST results >3.0 x ULN | 1 | 4 | 8

ADVERSE EVENTS:
Time Frame: Serious adverse event data collected through 288 weeks are presented.
Description: For the safety population, subjects were classified based on the highest dose of ambrisentan received at any time during the 2 prior studies (NCT00423748 or NCT00423202) or in the current extension study.
Groups:
- Ambrisentan 2.5 mg; Ambrisentan 5 mg; Ambrisentan 10 mg: Participants were classified based on the highest dose of ambrisentan received at any time during the 2 prior studies (NCT00423748 or NCT00423202) or in the current extension study. Study drug was taken once daily.
Arm/Group | Ambrisentan 2.5 mg | Ambrisentan 5 mg | Ambrisentan 10 mg
Serious Adverse Events (participants affected / at risk) | 26/43 | 76/146 | 103/194
Other Adverse Events (participants affected / at risk) | 36/43 | 131/146 | 190/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambrisentan 2.5 mg (N=43) | Ambrisentan 5 mg (N=146) | Ambrisentan 10 mg (N=194)
AV dissociation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 3 (3)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 4 (4) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Bone infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bone marrow depression (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (3) | 1 (1)
Bronchitis acute (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
CREST syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Catheter related complication (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (4) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 4 (4)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (2)
Dermoid cyst of ovary (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (3)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 4 (4)
Encephalitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Exercise capacity descreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fibroadenoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Heart and lung transplant (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 6 (8)
Hysteroscopy (Investigations) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Insulinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal functional disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Malignant soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Meningitis tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Mesenteric occlusion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Microlithiasis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 2 (2) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Neurosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Noncardiac chest pain (General disorders) | 0 (0) | 1 (1) | 4 (5)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 2 (2)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pacemaker complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Panic reaction (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Peritoneal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (7)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 5 (6) | 9 (13)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Polytraumatism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Postoperative infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 5 (5) | 2 (2)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 10 (12) | 33 (48)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Right ventricular failure (Cardiac disorders) | 6 (6) | 14 (18) | 34 (55)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Stevens Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 2 (2)
Sudden death (General disorders) | 0 (0) | 2 (2) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 3 (5)
Syncope (Nervous system disorders) | 3 (3) | 3 (3) | 5 (5)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5) | 1 (1)
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 2 (2)
Tachyarrhthmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Therapy regimen changed (Surgical and medical procedures) | 0 (0) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan 2.5 mg (N=43) | Ambrisentan 5 mg (N=146) | Ambrisentan 10 mg (N=194)
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 15
Abdominal pain (Gastrointestinal disorders) | 2 | 11 | 16
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6 | 21
Abnormal chest sound (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 10
Anaemia (Blood and lymphatic system disorders) | 6 | 19 | 26
Angina pectoris (Cardiac disorders) | 1 | 3 | 12
Anxiety (Psychiatric disorders) | 1 | 10 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 18 | 38
Asthenia (General disorders) | 3 | 8 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 11 | 36
Blood alkaline phosphatase increased (Investigations) | 4 | 3 | 6
Bronchitis (Infections and infestations) | 3 | 13 | 17
Bronchitis acute (Infections and infestations) | 3 | 4 | 7
Cardiac murmur (Investigations) | 2 | 4 | 10
Chest discomfort (General disorders) | 1 | 2 | 25
Chest pain (General disorders) | 1 | 6 | 15
Constipation (Gastrointestinal disorders) | 0 | 12 | 21
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 26 | 46
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 16
Cyanosis (Cardiac disorders) | 0 | 1 | 14
Depression (Psychiatric disorders) | 1 | 11 | 25
Diarrhoea (Gastrointestinal disorders) | 3 | 24 | 33
Dizziness (Nervous system disorders) | 3 | 15 | 47
Dyspepsia (Gastrointestinal disorders) | 1 | 7 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 13 | 29
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 4 | 19 | 35
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 31
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 11
Fatigue (General disorders) | 3 | 14 | 30
Fluid retention (Metabolism and nutrition disorders) | 0 | 2 | 10
Flushing (Vascular disorders) | 3 | 9 | 8
Gamma-glutamyltransferase increased (Investigations) | 4 | 9 | 13
Gastritis (Gastrointestinal disorders) | 1 | 13 | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 12
Headache (Nervous system disorders) | 1 | 34 | 61
Heart sounds abnormal (Investigations) | 0 | 4 | 13
Hepatomegaly (Hepatobiliary disorders) | 1 | 7 | 13
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 9 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 13 | 23
Hypotension (Vascular disorders) | 5 | 8 | 16
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 10
Influenza (Infections and infestations) | 5 | 13 | 22
Insomnia (Psychiatric disorders) | 2 | 13 | 23
International normalised ratio increased (Investigations) | 0 | 7 | 14
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1 | 12
Jugular vein distension (Vascular disorders) | 0 | 2 | 17
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 9 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 9 | 18
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 19 | 28
Nasopharyngitis (Infections and infestations) | 2 | 22 | 34
Nausea (Gastrointestinal disorders) | 3 | 12 | 38
Neck pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 10
Non-cardiac chest pain (General disorders) | 1 | 10 | 19
Oedema peripheal (General disorders) | 13 | 53 | 101
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 7 | 36
Palpitations (Cardiac disorders) | 3 | 12 | 35
Paraesthesia (Nervous system disorders) | 0 | 2 | 11
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 15
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 3 | 12
Pyrexia (General disorders) | 1 | 11 | 18
Rash (Skin and subcutaneous tissue disorders) | 1 | 5 | 12
Respiratory tract infection (Infections and infestations) | 2 | 6 | 24
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 12
Right ventricular failure (Cardiac disorders) | 4 | 15 | 20
Sinusitis (Infections and infestations) | 0 | 15 | 24
Syncope (Nervous system disorders) | 2 | 7 | 19
Tachycardia (Cardiac disorders) | 0 | 3 | 12
Upper respiratory tract infection (Infections and infestations) | 5 | 17 | 50
Urinary tract imfection (Infections and infestations) | 2 | 7 | 26
Vertigo (Ear and labyrinth disorders) | 0 | 5 | 19
Vomiting (Gastrointestinal disorders) | 0 | 7 | 23
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 7 | 12 | 32

LIMITATIONS AND CAVEATS:
Analysis included those not enrolling in this study but received AMB in 1 of the 2 parent studies. At Year 3, almost half of those randomized to 2.5 mg were titrated to 5 mg and 10 mg; a third starting at 5 mg were titrated to 10 mg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No